CLINICAL TRIAL: NCT03002870
Title: Characteristics of Patient Population With Endometriosis - A Prospective Database and BioBank
Brief Title: Characteristics of Patient Population With Endometriosis
Acronym: 20900
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Patrick Yeung Jr., MD, Principal Investigator, St. Louis University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20900
Record Dates: First submitted 2016-10-04; First posted 2016-12-26 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Endometriosis (Other): Patients whom pathology results post surgery document endometriosis
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Patients will receive questionnaires yearly to follow their QOL

SUMMARY:
The purpose of this study is to collect and analyze data on the characteristics of women who are seeking treatment for endometriosis, suspected endometriosis, pain and/or infertility as part of their standard medical care. Data collected will contribute to the development of guidelines for the surgical management of endometriosis. In addition, specimens will be collected for future testing regarding diagnosing, and/or staging of endometriosis, or suspected endometriosis, pain and infertility.

DETAILED DESCRIPTION:
Patients seen at Saint Louis University Center for Endometriosis (which has offices locations at St. Mary's, St. Luke's and the SLU-UMG clinic - all of which are in the SLU Epic system), and operated on for endometriosis, suspected endometriosis, pain and/or infertility at St. Mary's hospital (only).

A preoperative questionnaire will be provided to the subject. Questions from the survey include information on baseline demographics, severity and type of pain, and previous medical and surgical history. Operative data will also be collected and analyzed.

A post-operative questionnaire will be administered to the participants at 6 months, and then at regular yearly intervals after the surgery by a secure on-line process using the RedCap software. Improvement in quality of life and pain scores will be analyzed.

Specimens will also be collected and stored for future testing regarding diagnosing, and/or staging of endometriosis, suspected endometriosis, pain and infertility.

ELIGIBILITY:
Inclusion Criteria:

* Female patients
* 13-55 years of age
* Anyone seen at the Center for Endometriosis

Exclusion Criteria:

* Prior bilateral salpingo-oophorectomy
* post natural menopause
* Significant mental or chronic systemic illness that might confound pain assessment or the inability to complete the study.

Ages: 13 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1100 (Actual)
Dates: Start 2016-09; Primary Completion 2024-09-04 (Actual); Study Completion 2024-09-04 (Actual)

PRIMARY OUTCOMES:
Quality of life, pain and fertility | every 12 months
  (QOL) endometriosis health profile (EHP-5)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Yeung, MD, Principal Investigator — St. Louis University
Locations (1):
- Saint Louis University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No